CLINICAL TRIAL: NCT07266584
Title: Restoration of Central Vision With the PRIMA Products in Patients With Photoreceptor Degeneration
Brief Title: Restoration of Central Vision With PRIMA in Patients With Photoreceptor Degeneration
Acronym: PRIMAlia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-PRIMA-AUS
Record Dates: First submitted 2025-11-19; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Stargardt Disease; Retinitis Pigmentosa (RP); Inherited Retinal Degeneration
MeSH Terms: conditions — Stargardt Disease; Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRIMA Products (Experimental)
  Interventions: Device: PRIMA Products

INTERVENTIONS:
Device: PRIMA Products — Implantation of PRIMA, Vision training, follow up

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of the PRIMA Products in participants with inherited retinal degeneration affecting the macula (including but not limited to Stargardt disease, and Retinitis Pigmentosa).

Eligible participants will be implanted with the PRIMA Stim implant. The participants will be assessed with various visual function and functional vision tests at defined timepoints throughout the clinical investigation with the PRIMA Products. The purpose of this study is to gather enough clinical data to support the clinical evaluation required for the continuous development to improve the PRIMA Products.

DETAILED DESCRIPTION:
Science has developed the PRIMA Products, which are designed to restore limited visual perception in severely sight-impaired persons with a functional optic nerve and retinal ganglion cell layers who have lost their central vision due to the degeneration of photoreceptor cells.

The PRIMA Products have been tested successfully in 38 patients with Geographic Atrophy. PRIMA was found to be both safe and effective in this population. This exploratory study is to investigate whether patients with inherited retinal degeneration affecting the macula can also benefit from PRIMA.

The objective of this study is to evaluate the efficacy and safety of the PRIMA Products in participants with inherited retinal degeneration, affecting the macula and resulting in photoreceptor degeneration, including Stargardt disease and retinitis pigmentosa. The investigation is sponsored by Science Corporation Australia.

ELIGIBILITY:
Inclusion Criteria:

1. Is 18 years or older at the date of inclusion;
2. Has a confirmed diagnosis of inherited retinal degeneration with the macula affected in both eyes;
3. The study eye has best corrected visual acuity of logMAR 1.2 (20/320) or worse as measured by ETDRS test;
4. Has an atrophic patch in the study eye including the fovea of at least the implant size (>4.5 mm2 and >2.4 mm in minimum diameter);
5. Understands the constraints of the study and accepts to present for all scheduled follow-up visits;
6. Signed the informed consent.

Exclusion Criteria:

1. 1. Has cataract in the study eye (with LOCS III scale NO, NC, C or P>1); (these patients will need to have cataract surgery performed prior to completion of baseline testing; all other patients will get IOL replacement during the PRIMA Stim implantation);
2. Underwent intraocular lens implantation in the study eye within the last month prior to enrolment (this corresponds to 4 weeks or 28 days) ;
3. Has an implanted IOL in the study eye and a refraction of the study eye outside of -4D; +4D limit (this criterion is not relevant for phakic eyes)
4. Has a highly myopic study eye (>26 mm AP);
5. Has no light perception in either eye;
6. Has a history of documented choroidal neovascularization in either eye;
7. Has any signs of exudative AMD including exudative AMD with detachment of retinal pigment epithelium in the central visual field of the study eye;
8. Has an implanted telescope in one eye;
9. Has a black IOL in the study eye;
10. Has any disease (other than study allowed diseases) or condition that affects retinal function of the study eye or the visual system (e.g., central retinal artery/vein occlusion, end-stage diabetic retinopathy, Proliferative Diabetic Retinopathy (PDR), diabetic macular oedema (DME), severe Non-Proliferative Diabetic Retinopathy (NPDR), retinal detachment, infectious or inflammatory retinal disease, severe glaucoma, optic neuropathy, etc.) ;
11. Has any disease or condition that prevents adequate examination (including Optical Coherence Tomography (OCT)) of the study eye including but not limited to media opacities that cannot be resolved prior to implantation. Note, that this criterion is also important for the function of the implant;
12. Has a corneal endothelial cell count of less than 1000 cells/mm² in the study eye;
13. Suffers from nystagmus or other ocular motility disorders;
14. Has any disease or condition that precludes the understanding or communication of the informed consent, study requirements or test protocols (e.g., deafness, severe multiple sclerosis, amyotrophic lateral sclerosis, severe neuritis, etc.);
15. Has uncontrolled epileptic seizures;
16. Has a known sensitivity to the contact materials of the implant (iridium oxide, silicon-carbide and titanium);
17. Has a known allergy to anaesthetic drugs;
18. Presents with hypotonia in the study eye (<8 mmHg);
19. Presents with hypertonia in the study eye (>23 mmHg with treatment);
20. Has active cancer or a history of intraocular, optic nerve or brain cancer and metastasis;
21. Is an immune-suppressed participant (e.g., due to HIV positive diagnosis, etc.);
22. Is a known carrier of multi-resistant microorganisms;
23. Is receiving anticoagulation therapy that cannot be adapted to allow eye surgery;
24. Is participating in another investigational drug or device study that may interfere with the PRIMAlia study;
25. Has a history of chronic or recurrent infection or inflammation that would preclude participation in the study;
26. Has significant recurrent or chronic inflammations or infections. Specifically, patients with the following disorders are excluded:

    * Severe chronic and consuming diseases that frequently associated with infection (e.g. Crohn disease, Whipple's disease);
    * Active inflammation in the area of the eye (e.g. herpes of cornea and/or conjunctiva, recurrent blepharoconjunctivitis, hordeolum, chalazion);
27. Has a severe psychological disorder;
28. Does not have the mental capacity to legally sign the informed consent;
29. Has severe renal, cardiac, hepatic, etc. organ diseases (ASA IV or worse);
30. Has head dimensions that are incompatible with the PRIMA Companion glasses;
31. Has too high and/or unrealistic expectations (e.g., believes that a benefit is guaranteed or expects normal vision after surgery).
32. Physical constraints making use of PRIMA or rehabilitation impossible
33. Participant who, in the opinion of the investigator, is not suitable for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with an improvement of visual acuity | 12 months
  Proportion of participants with an improvement of visual acuity of logMAR 0.2 or more
Number and severity of device and procedure related serious adverse events | 12 months
  Number and severity of device and procedure related serious adverse events

SECONDARY OUTCOMES:
Proportion of participants with an improvement of visual acuity | 6, 24 and 36 months
  Proportion of participants with an improvement of visual acuity of logMAR 0.2 or more
Mean improvement in visual acuity | 6, 12, 24 and 36 months
  Mean improvement in visual acuity measured by ETDRS (extended by the Berkeley Rudimentary Vision Test)
Mean improvement in the reading test | 12, 24 and 36 months
  Mean improvement in the reading test
Number and severity of procedure and device related adverse events throughout the study | up to 36 months
  Number and severity of procedure and device related adverse events throughout the study
Change of natural visual acuity | up to 36 months
  Change of natural visual acuity from baseline without the PRIMA Companion glasses measured by ETDRS (extended by the Berkeley Rudimentary Vision Test)

CONTACTS AND LOCATIONS:
Locations (1):
- Sydney Eye Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Science Corporation — https://science.xyz/